CLINICAL TRIAL: NCT04021524
Title: Randomized Trial of Hibiclens vs Benzoyl Peroxide Soap for Surgical Preparation
Brief Title: BPO vs Hibiclens Soap for Surgical Preparation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Frederick Matsen, Professor and Chairman, School of Medicine: Orthopaedics and Sports Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00005028
Record Dates: First submitted 2019-07-01; First posted 2019-07-16 (Actual); Results first posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2021-12

CONDITIONS: Propionibacterium Acnes
MeSH Terms: interventions — Benzoyl Peroxide; Receptors, Catecholamine; chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hibiclens Soap (Active Comparator)
  Interventions: Drug: Chlorhexidine Gluconate
- BPO Soap (Experimental)
  Interventions: Drug: Benzoyl Peroxide 10% Bar

INTERVENTIONS:
Drug: Benzoyl Peroxide 10% Bar — Patients will wash with Benzoyl Peroxide 10% Bar
  Arms: BPO Soap
Drug: Chlorhexidine Gluconate — Patients will wash with Chlorhexidine Gluconate
  Arms: Hibiclens Soap

SUMMARY:
This is a randomized trial of benzoyl peroxide soap versus Hibiclens soap for surgical preparation. The objective is to determine whether benzoyl peroxide soap, commonly available in drug stores for over-the-counter acne treatment, is as or more effective than the standard surgical preoperative soap, Hibiclens soap (chlorhexidine gluconate), in reducing loads of Propionibacteria (Propi) on or under the skin of patients prior to shoulder arthroplasty (joint replacement).

ELIGIBILITY:
Inclusion Criteria:

* Male subjects
* Subjects scheduled for elective shoulder arthroplasty at the University of Washington Medical Center
* Subjects between ages 18-89

Exclusion Criteria:

* Subjects who self-report very sensitive skin
* Subjects who are sensitive to benzoyl peroxide
* Subjects who are allergic to chlorhexidine
* Subjects who had recent prior use of antibiotics (or expect to use them prior to surgery)
* Subjects who had recent use of acne treatment
* Subjects who are not fluent in English.

Ages: 18 Years to 89 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2021-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Matsen, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hibiclens Soap | BPO Soap
Started | 25 | 25
Completed | 25 | 24
Not Completed | 0 | 1
Not completed — Change in surgical intervention | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hibiclens Soap | BPO Soap | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (11.1) | 63.4 (11.1) | 64.4 (11.0)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 25 | 24 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 25 | 22 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Body Mass Index [Median (Standard Deviation); unit: kg/m^2] | 28.8 (6.1) | 30.3 (5.9) | 29.5 (6.0)
Prior Shoulder Surgery [Count of Participants; unit: Participants] | 16 | 4 | 20
ASA Classification [Count of Participants; unit: Participants] — I - A normal healthy patient ; II - A patient with mild systemic disease ; III - A patient with severe systemic disease ; IV - A patient with severe systemic disease that is a constant threat to life
  Participants
    I | 5 | 0 | 5
    II | 14 | 17 | 31
    III | 6 | 7 | 13
    IV | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With a Positive Propionibacteria Swabs on Day of Surgery After At-Home Washes With Benzoyl Peroxide or Chlorhexidine Gluconate
Description: Patients were randomly assigned to use either benzoyl peroxide soap or Hibiclens soap (chlorhexidine gluconate) at home the night before and the morning of surgery. On the day of surgery the patients' skin and incisions were swabbed in the operating room prior to shoulder arthroplasty. Specimens were held for 21 days.
Time Frame: Day of Surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Hibiclens Soap | BPO Soap
Number analyzed (Participants) | 25 | 24
Participants
  Skin Surface Positive Swab | 25 | 24
  Dermal Edge Positive Swab | 14 | 11

2. Primary Outcome: Number of Quadrants on Culture Plate of Propionibacteria Growth - Specimens Taken Day of Surgery After At-Home Washes With Benzoyl Peroxide or Chlorhexidine Gluconate
Description: This outcome measures the load of Propionibacteria on the skin and incision of participants in the operating room prior to shoulder arthroplasty when patients were randomly assigned to use either benzoyl peroxide soap or Hibiclens soap (chlorhexidine gluconate) at home the night before and the morning of surgery. The Propionibacteria load was quantified based on the growth of bacteria on the agar plate using a quadrant system. Quantitative specimen Propionibacteria values (SpCuVs) were assigned as following: "no growth"= 0, "broth only"= 0.1, "one colony only"= 0.1, and 1 quadrant growth = 1, 2 quadrant growth = 2, 3 quadrant growth = 3, and 4 quadrant growth = 4. Samples were taken on the day of surgery and the cultures were held for 21 days.
Time Frame: Day of Surgery
Measure: Mean (Standard Deviation); unit: SpCuV
Arm/Group | Hibiclens Soap | BPO Soap
Number analyzed (Participants) | 25 | 24
SpCuV
  Skin Surface SpCuV | 1.6 (1.1) | 1.5 (1.4)
  Dermal Edge SpCuV | 0.8 (1.0) | 0.8 (1.4)

ADVERSE EVENTS:
Time Frame: Day of surgery
Description: Cultures were taken on the day of surgery and held for 21 days. Adverse events were assessed after the culture results were finalized.
Arm/Group | Hibiclens Soap | BPO Soap
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 0/25 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/24/NCT04021524/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-07): https://cdn.clinicaltrials.gov/large-docs/24/NCT04021524/ICF_001.pdf